CLINICAL TRIAL: NCT06253923
Title: Multicenter, Double-blind, Randomized, Placebo Controlled, Study to Assess the Safety of Amantadine Hydrochloride (HCl) Intravenous (IV) Solution (MR-301), in Patients With Severe Traumatic Brain Injury (TBI).
Brief Title: Study to Assess the Safety of Amantadine Hydrochloride (HCl) Intravenous (IV) Solution (MR-301) in Patients With Severe Traumatic Brain Injury (TBI).
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SHINKEI Therapeutics, Inc (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR-301-T-001
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MR-301 (Active Comparator): On first day, patient will receive MR-301 at 100 mg intravenous infusion BID. On second day, the dose is elevated to 150 mg intravenous infusion BID.
  On third day, the dose is further elevated to 200 mg intravenous infusion BID and maintained up to Day 21
  Interventions: Drug: Amantadine Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine Hydrochloride — MR-301 is an I.V. formulation for the treatment of TBI. The active ingredient is amantadine hydrochloride (HCl).
  Arms: MR-301
Drug: Placebo — The placebo for this study is 0.9% Sodium Chloride IV Solution.
  Arms: Placebo

SUMMARY:
The main goal of this clinical trial is to check if the treatment is safe and well-tolerated. Researchers will compare the MR-301 active drug group with the placebo group to evaluate the safety and tolerability of the drug. Other measurements include assessing the patient's overall outcome, neurological responses, time spent in the intensive care unit, time in the hospital, and mortality. Participants will receive either MR-301 BID IV dosing or a matching placebo for a total of 3 weeks.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled study of MR-301 administered BID IV in patients with severe TBI.

Participant: 45 patients with severe TBI who maintain GCS scores 3-8 both inclusive.

Intervention: Mr-301 or placebo will be administered intravenously BID for upto 3 weeks.

Primary Outcome: Safety and Tolerability of MR-301

Secondary Outcome: GOS-E, CRS-R, DRS, FOUR score, time to ICU discharge, time to hospital discharge and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years.
2. Patients with TBI confirmed by CT scan or MRI
3. Patient have sustained a trauma between 72 hours to 1 week
4. Patient with Abbreviated Injury Score (AIS) ≤ 2.
5. Patients must be admitted to an acute care setting no less than 2 days prior to randomization.
6. Glasgow Coma Score of 3 to 8, inclusive.
7. Patients must be unable to consistently follow commands or to engage in functional communication, as assessed by the score on the CRS-R.
8. Patients have at least one reactive pupil.
9. Must have a Legally Authorized Representative (LAR) able to provide consent for the trial.
10. Patient must have stable vitals ---Intracranial pressure ICP Value is at discretion of investigator), systolic blood pressure (SBP>90 mmHg) partial pressure of oxygen (PaO2 > 60 mmHg)].

Exclusion Criteria:

1. Life expectancy of less than 24 hours.
2. Patient has any spinal cord injury.
3. Patient has a penetrating head injury.
4. Patient has bilaterally fixed dilated pupils
5. Patients with history of any medical or psychiatric disorder, or any severe concomitant disease that would, in the opinion of the Investigator, interfere with clinical assessment.
6. Patient has poorly controlled seizure more than one per month.
7. Prior history of status epilepticus
8. Prior treatment with or a sensitivity to amantadine HCl or amantadine.
9. Patient has screening lab measurements outside the normal range

   1. Absolute neutrophil count (ANC): ≤ 1.5 x 109/L
   2. Hemoglobin ≤ 8 g/dL or active bleeding requiring ongoing transfusions.
   3. Platelets ≤ 80 x 109/L or active bleeding requiring ongoing transfusions.
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) or total bilirubin (unless isolated Gilbert's syndrome) ≥ 2x the upper limit of normal (ULN)
   5. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2
10. Patient has received treatment with an investigational drug, CNS stimulant or dopamine antagonist/agonist within 4 weeks.
11. Patient has a history of NYHA Class 3 or Class 4 Congestive Heart Failure within the last 5 years.
12. Females who are nursing, pregnant, or planning to become pregnant
13. any other clinically significant medical condition as determined by the Investigator, that may unfavorably alter the risk benefit of study participation.
14. Patient has prolonged QT interval.
15. Treatment with a systemic anticholinergic medication within 1 week prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Frequency, severity, and type of adverse events and serious adverse events between active treatment and placebo groups | Day 1 to Day 35
  Safety and tolerability will be compared between active treatment and placebo groups.

SECONDARY OUTCOMES:
Change from baseline in Glasgow Outcome Scale-Extended | Day 21 and Day 35
Change from baseline in Disability Rating Scale (DRS) scale | Day 5, Day 10, Day 15, Day 21
Change from baseline in Coma Recovery Scale - Revised | Day 5, Day 10, Day 15, Day 21
Change from baseline in Full Outline of UnResponsiveness (FOUR) score | every day up to Day 21
Time to intensive care unit (ICU) discharge to hospital floor | up to day 21
Time to hospital discharge from randomization | up to day 21
Mortality assessment at end of treatment period | Day 21
Mortality assessment at end of study period (Day 35). | Day 35

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Los Angeles General Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UF Health Heart and Vascular Hospital, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Maine Medical Center, Portland, Maine
  - Wayne State University, Detroit, Michigan
  - Barnes Jewish Hospital, St Louis, Missouri
  - Hackensack Meridian Health Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Department of Neurology, Duke University School of Medicine, Durham, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - McGovern Medical School, University of Texas Health Science Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No